CLINICAL TRIAL: NCT07070869
Title: SPAMLO-3.0 : Having Fun Shedding Light on Darkness
Brief Title: SPAMLO-3.0 : Having Fun Shedding Light on Darkness, a Playful Approach to Reduce Anxiety in Palliative Care
Acronym: SPAMLO 3 0
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024_CHSB_SPAMLO-3.0; 2024-A02381-46 (Other: ID RCB)
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Palliative Care; Serious Games; Anxiety
Keywords: anxiety; serious game; palliative care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Standard care by the healthcare team and participation in the serious game "SPAMLO-3.0."
  Interventions: Behavioral: Serious game
- Control group (No Intervention): Standard care provided by the mobile palliative care team, according to the usual practices of the healthcare team.

INTERVENTIONS:
Behavioral: Serious game — Participation in the serious game "SPAMLO-3.0."
  Arms: Intervention group

SUMMARY:
End-of-life care is often accompanied by anxiety-not only for patients in palliative care, but also for their loved ones and the healthcare professionals supporting them. This anxiety may stem from a fear of death, loss of functional abilities, or a worsening of symptoms as the illness progresses.

It contributes to emotional, psychological, and physical suffering, ultimately diminishing patients' quality of life. Most data on palliative care focus on cancer patients, among whom anxiety prevalence varies greatly, but may affect more than 70% of individuals.

Currently, anxiety in palliative care patients is managed through non-pharmacological approaches (such as environmental modifications and relaxation techniques) and/or pharmacological treatments (including antidepressants, neuroleptics, and anxiolytics).

The investigators recently developed the serious game SPAMLO with the aim to present and raise awareness about palliative care. The educational scenario was built around three settings: the hospital, the home, and the nursing home (EHPAD). The participant will follow Vito, a virtual character, whose sister is receiving palliative care. Vito will explore the different types of support available, starting at the hospital. He will learn about what a collegial discussion is, the Clayes-Léonetti law, advance directives, the trusted person, as well as the specificities of pediatrics. Through home hospitalization, Vito will discover palliative care outside the hospital setting, including home adaptations with appropriate equipment and the various available support services. Finally, Vito will visit the nursing home, where topics such as oral care, respecting the patient's choices, and the importance of preserving them will be addressed.

Thanks to its playful approach and the knowledge gained, this game could help reduce anxiety in palliative care patients through non-pharmacological means. This research project has beeen co-designed with a JALMALV volunteer (Accompany life until death - french association).

DETAILED DESCRIPTION:
Participants will be randomly assigned to two groups (at a 1:1 ratio):

Control group: standard care provided by the mobile palliative care team, according to the usual practices of the healthcare team.

Intervention group: standard care by the healthcare team plus participation in the serious game "SPAMLO-3.0."

Participants will have 7 days to complete the game (multiple sessions allowed). Participant's anxiety and secondary outcomes will be measured on Day 15 to assess the primary endpoint.

A second evaluation is planned on day 30 for secondary endpoints. This second assessment will allow participants time to reflect following their participation in the serious game, potentially encouraging the designation of a trusted person and the drafting of advance directives.

Demographic, clinical, therapeutic characteristics, and questionnaires will be collected at inclusion, Day 15, and Day30. The study duration for each participant is 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant for whom no curative treatment is proposed, who is either discharged home or hospitalized in palliative care
* Life expectancy presumed to be greater than one month
* No cognitive impairments, according to the healthcare team's assessment
* Participantt has given free and informed consent
* Participant affiliated with a social security system
* The participant owns a computer, tablet, or smartphone with an internet connection and agrees to participate in the serious game SPAMLO-3.0.

Exclusion Criteria:

* Participant who is demented, confused, or in a coma
* Fatigability, according to the healthcare team's assessment
* Visually or hearing impaired participant, according to the healthcare team's assessment
* No inclusion of persons targeted by Articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the Public Health Code (e.g., minors, legally protected adults, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depresion Scale | Day 0, Day 15 and Day 30
  Questionnaire completed by the participant. It consists of 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and the other seven to the depressive dimension (total D), thus allowing for the calculation of two scores (maximum score for each = 21).
  The scores for each of the Anxiety and Depression subscales are interpreted as follows:
  0 to 7: no signs of anxiety and/or depressive disorders. 8 to 10: borderline or doubtful symptomatology. 11 to 21: confirmed anxiety and/or depressive disorders of varying severity.

SECONDARY OUTCOMES:
Acceptability of the serious game through a Likert questionnaire | Day 30
  Likert questionnaire completed by the participant
Number of participants who completed the serious game. | Through study completion, an average of 20 months
  Data obtained by the coordinating investigator
French System Usability Scale | Through study completion, an average of 20 months
  Healthcare team's perception of the use of the serious game. The questionnaire includes ten items, each formulated as a statement. For each statement, the user is asked to indicate their level of agreement or disagreement using a 5-point Likert scale (1 = Strongly disagree; 5 = Strongly agree). If the user is unsure how to respond to an item, they are encouraged to answer anyway by selecting the middle point of the scale (score 3).
McGill Quality of Life Questionnaire | Day 0, Day 15 and Day 30
  Completed by the participant. It is a 17-item multidimensional tool designed to measure physical well-being, physical symptoms, psychological symptoms, existential well-being and support, as well as overall quality of life. The scores for each domain are calculated separately.
Insomnia Severity Index | Day 0 and Day 30
  Completed by the participant. The first item assesses the intensity of insomnia complaints separately for difficulty falling asleep, maintaining sleep, and early awakening. One item evaluates the subject's overall satisfaction with their sleep, and another item assesses concerns regarding insomnia. Finally, two items evaluate the impact on daily life activities. Each item is rated by the patient from 0 to 4.The total score ranges from 0 to 28.
  * between 0 and 7 indicates the absence of clinically significant insomnia complaints,
  * between 8 and 14 indicates subclinical (mild) insomnia complaints,
  * between 15 and 21 indicates clinically significant (moderate) insomnia complaints,
  * between 22 and 28 indicates severe insomnia complaints.
Palliative Performance Scale | Day 0, Day 15 and Day 30
  Completed by investigators. This is an 11-point scale used to measure a patient's performance in 10% increments, with 100% representing health and 0% representing death. The scale is based on five observable parameters: mobility, activity level, independence in personal care, feeding, and level of consciousness.
Visual analog scale | Day 0, Day 15 and Day 30
  Evaluated by the participant.
  This scale measures pain intensity on a scale from 0 to 10. The correspondence between VAS (Visual Analog Scale) levels and pain intensity is as follows:
  * between 1 and 3: mild pain intensity
  * between 3 and 5: moderate pain intensity
  * between 5 and 7: severe pain intensity
  * above 7: very severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie LOUICHE, Principal Investigator — Centre Hospitalier de Saint-Brieuc - Paimpol - Tréguier
Locations (1):
- Centre Hospitalier de Saint-Brieuc - Paimpol - Tréguier, Saint-Brieuc, France

IPD SHARING:
Plan to Share IPD: Undecided